CLINICAL TRIAL: NCT06248021
Title: Effectiveness of Ecological Footprint Awareness Program in 60-72 Months Children: A Randomized Controlled Study
Brief Title: Ecological Footprint Awareness Program in 60-72 Months Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Ayse Sezer Balci, Assistant Professor, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ERSOYU-SBF-ASB-01
Record Dates: First submitted 2024-01-24; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Program, Communication
Keywords: environment; ecology; awareness; child
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This study was conducted using a cluster randomized controlled pretest-posttest experimental design. It was carried out in four kindergartens located in a city center between April and June 2023. Two of the kindergartens were assigned to the intervention group while the other two were assigned to the control group. Data was collected using the Ecological Footprint Awareness Scale for Children (EFAS-C). The training program was conducted with the children in the intervention group for four weeks, with a 40-minute session each week. The program covered one topic each week, which included waste management, water and energy use, food consumption, and transportation.
Who Masked: Participant, Investigator
Masking Description: The researcher responsible for the study identified the children who were assigned to the intervention and control groups. This person was not involved in the implementation of the study to ensure that measurement bias was controlled. To avoid detection bias, statistical bias, and reporting bias, a third researcher, who did not know which children were in the intervention and control groups, was responsible for coding and analyzing the research data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ecological Footprint Awareness Program Group (Experimental): The program was conducted for four weeks, one day each week, for 40 minutes. Each week, a different topic was addressed such as waste evaluation, water and energy usage, food consumption, and transportation. The program was created in line with expert opinions and literature.
  Interventions: Behavioral: Ecological Footprint Awareness Program
- Control Group (No Intervention): No intervention was applied to the group

INTERVENTIONS:
Behavioral: Ecological Footprint Awareness Program — The program was conducted for four weeks, one day each week, for 40 minutes. Each week, a different topic was addressed such as waste evaluation, water and energy usage, food consumption, and transportation. The program was created in line with expert opinions and literature. The sessions were based on the principles of the Social Cognitive Learning Theory, developed by Bandura, which includes mutual determinism, symbolization, anticipatory capacity, vicarious learning, self-regulation capacity, and self-judgment capacity. During each session, various techniques such as animation, drawing, storytelling, memory cards, and games were employed. To ensure the program's content was appropriate for children's development, the opinions of two experts from the child development department of the university were obtained.
  Arms: Ecological Footprint Awareness Program Group

SUMMARY:
This study aimed to evaluate the effectiveness of an ecological footprint awareness training program for children aged 60-72 months.

DETAILED DESCRIPTION:
This study was conducted using a cluster randomized controlled pretest-posttest experimental design. It was carried out in four kindergartens located in a city center between April and June 2023. Two of the kindergartens were assigned to the intervention group while the other two were assigned to the control group. Data was collected using the Ecological Footprint Awareness Scale for Children (EFAS-C). The training program was conducted with the children in the intervention group for four weeks, with a 40-minute session each week. The program covered one topic each week, which included waste management, water and energy use, food consumption, and transportation. The data was analyzed using descriptive statistics, paired groups t-test, and independent groups t-test, with a 95% confidence interval and p<.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in the schools where the study was conducted
* Approved by their family to participate in the study,
* 60-72 months old

Exclusion Criteria:

* participation in less than 2/3 of the intervention protocol

Ages: 60 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Ecological Footprint Awareness Scale for 60-72 Month-old Children scores | four weeks
  ıt contains five themes, including 'Water and energy use,' 'Waste utilization,' 'Food consumption,' and 'Transportation'. It contains a total of 19 items, which are asked through a game and story structure. he scale is divided into two sections: a game section and a story section. In the game section, children are shown pictures and asked how the characters should behave. In the story section, children are told a story and asked which character is behaving in an environmentally friendly way. Children who answer correctly receive a score of "1", while those who answer incorrectly receive a score of "0". The total score is used to measure environmental awareness. The KR-20 coefficient for internal consistency reliability of the EKAY-O was calculated as 0.66.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided